CLINICAL TRIAL: NCT01699893
Title: Genetic & Environmental Determinants Of Immune Phenotype Variance: Establishing A Path Towards Personalized Medicine
Acronym: LabExMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2012-A00238-35
Record Dates: First submitted 2012-09-21; First posted 2012-10-04 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Individuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- unique arm (Experimental): * At V0: 1500 will be screened
  * At V1: 1000 subjects will be performed following samples: blood, nasal swab,stool. 500 subjects among 1000 will be performed one additional sample (Skin Biopsy)
  * At V2: only the 500 subjects having performing the skin biopsy at V1 will come at V2 to perform blood, nasal swab and stool samples
  Interventions: Other: unique arm

INTERVENTIONS:
Other: unique arm — blood, nasal swab, skin biopsy, stool samples

SUMMARY:
The purpose of this study is to assess the determinants of immunologic variance within the general healthy population.

DETAILED DESCRIPTION:
Susceptibility to infections, disease severity, and response to medical therapies and vaccines are highly variable from one individual to another. While the question of variance in human populations continues to be a focal point of scientific research, medical practices and public health policies typically take a 'one size fits all' model to disease management and drug development.

Individual heterogeneity in the immune response can have an enormous impact on the likelihood to respond to therapy or the development of side effects secondary to vaccine administration. Because of the complexity of immune responses in the individual and within the population, it has not been possible thus far to define the parameters (genetic or environmental) that constitute a healthy immune system and its natural occurring variability.

Efforts to restore the 'personal' in medical care are the current challenge, and the driving vision of the project, to which the current study belongs.

In order to realize the promise of personalized medicine, an in-depth understanding of the determinants of heterogeneity in host response to stress is required.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects considered as healthy by the investigator based on medical history, clinical examination, laboratory results and ECG (blood sampling for laboratory assessments and ECG should be done at V0 and only after signed informed consent).
2. Subjects who, according to the investigator, can and will comply with the requirements of the protocol and are available for all scheduled visits at the investigational site.
3. Healthy male or female aged between 20 and 69 (included) years
4. Metropolitan French origin for 3 generations 5)18.5 ≤BMI ≤ 32 kg/m² (Appendix 18.6)

6)Ability to give their informed consent in writing 7)Must understand spoken and written French 8)Affiliated to the French social security or assimilated regimens 9)Registered on the French "Fichier des Volontaires se prêtant à la Recherche Biomédicale (VRB)"

Exclusion Criteria:

1. Subjects who can not participate according to their status on the registry mentioned at Art L. 1121-16 of the French Public Health Code
2. Participation in another clinical study in the last 3 months in which the subject has been exposed to an investigational product (pharmaceutical product or placebo or medical device) or concurrent participation in another clinical study during the study period
3. Relatedness to previously recruited individuals in the study cohort
4. Travel in (sub-)tropical countries within the last 3 months
5. For women: pregnant or breastfeeding or intending to become pregnant or peri-menopausal*

   * Peri-menopausal women as defined by menstrual irregularity: either a change in the menstrual cycle length of more than seven days (early perimenopause) or two or more missed periods with an interval of 60 days or more between periods (late perimenopause) (Stages of Reproductive Aging Workshop, STRAW)(11)
6. Any physical exercise within the last 8 hours before inclusion (V1) and before (V2)
7. Subjects following a special diet for medical reasons as prescribed by a GP or dietician (e.g. calorie restricted or weight-loss diet for significant overweight, cholesterol lowering diet or subjects suffering from any clinically diagnosed food allergy or intolerance)
8. Alcohol abuse (more than 50 g of pure ethanol per day: for example, more than 4 x 150 mL glasses of wine, more than 4 x 250 mL glasses of beer, more than 4 x 40 mL glasses of high alcohol content drinks)
9. Illicit drug use or substance abuse within 3 months prior to inclusion
10. Presence of evidence of neurological or psychiatric diagnoses which, although stable, are deemed by the investigator to render the potential subject unable/unlikely to participate in the study satisfactorily.
11. Severe/chronic/recurrent pathological conditions,
12. Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within the 6 months prior to the inclusion. For corticosteroids, this will mean a dose equivalent to 20 mg/day of prednisone or equivalent for > 2 weeks (inhaled and topical steroids allowed)
13. Chronic administration of NSAIDs, including aspirin: prolonged intake (> 2 weeks) within 6 months before study or any intake within the 7 days preceding skin biopsy [exception for low dose aspirin: maximum 250mg/daily, see 8.1]
14. Receipt of any vaccination 3 months before the inclusion or planning to receive any vaccination during the study
15. Receipt of blood products or immunoglobulins within 3 months prior the inclusion or planning to receive blood products or immunoglobulins during the study
16. Hemoglobin measurement less than 10.0 g/dL for women and less than 11.5 g/dL for men
17. Platelet count less than 120.000/mm3
18. ALAT and/or ASAT > 3 times the upper limit of the norm (ULN)
19. Allergy to lidocaine

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1012 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Measurement of cytokine/chemokine stimulated by 40 pattern-recognition receptors agonists (PRR agonists) or immune stimulators. | V2 (28days after V1)

SECONDARY OUTCOMES:
Determination of genotype-to-phenotype associations at a mechanistic level | 4 days after V0

CONTACTS AND LOCATIONS:
Overall Officials: Matthew ALBERT, Study Chair — Institut Pasteur / Inserm; Lluis QUINTANA-MURCI, Study Chair — Institut Pasteur / CNRS; Nicolas FAUCHOUX, Principal Investigator — Biotrial Rennes
Locations (1):
- BIOTRIAL, Rennes, France

REFERENCES:
- [Derived] Scepanovic P, Hodel F, Mondot S, Partula V, Byrd A, Hammer C, Alanio C, Bergstedt J, Patin E, Touvier M, Lantz O, Albert ML, Duffy D, Quintana-Murci L, Fellay J; Milieu Interieur Consortium. A comprehensive assessment of demographic, environmental, and host genetic associations with gut microbiome diversity in healthy individuals. Microbiome. 2019 Sep 13;7(1):130. doi: 10.1186/s40168-019-0747-x. PMID 31519223
- [Derived] Partula V, Mondot S, Torres MJ, Kesse-Guyot E, Deschasaux M, Assmann K, Latino-Martel P, Buscail C, Julia C, Galan P, Hercberg S, Rouilly V, Thomas S, Quintana-Murci L, Albert ML, Duffy D, Lantz O, Touvier M; Milieu Interieur Consortium. Associations between usual diet and gut microbiota composition: results from the Milieu Interieur cross-sectional study. Am J Clin Nutr. 2019 May 1;109(5):1472-1483. doi: 10.1093/ajcn/nqz029. PMID 31051503
- [Derived] Scepanovic P, Alanio C, Hammer C, Hodel F, Bergstedt J, Patin E, Thorball CW, Chaturvedi N, Charbit B, Abel L, Quintana-Murci L, Duffy D, Albert ML, Fellay J; Milieu Interieur Consortium. Human genetic variants and age are the strongest predictors of humoral immune responses to common pathogens and vaccines. Genome Med. 2018 Jul 27;10(1):59. doi: 10.1186/s13073-018-0568-8. PMID 30053915